CLINICAL TRIAL: NCT00473863
Title: Coronary Computed Tomographic Angiography in Emergency Department Chest Pain Patients at Intermediate Risk of Acute Coronary Syndrome
Acronym: CCTA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver General Hospital (Other)
Collaborators: University of British Columbia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: H07-00742
Record Dates: First submitted 2007-05-15; First posted 2007-05-16 (Estimated); Last update posted 2007-11-20 (Estimated); Status verified 2007-11

CONDITIONS: Acute Coronary Syndrome; Acute Myocardial Infarction; Unstable Angina; Coronary Disease; Coronary Stenosis
Keywords: Acute coronary syndrome; Acute myocardial infarction; Unstable angina; Coronary computed tomographic angiography; Coronary Angiography; Tomography, X-Ray Computed; Tomography, Spiral Computed
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Coronary Disease; Coronary Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- intervention (Experimental): Receives CCTA
  Interventions: Procedure: Coronary Computed Tomographic Angiography
- Control (No Intervention)

INTERVENTIONS:
Procedure: Coronary Computed Tomographic Angiography — CCTA will be performed
  Arms: intervention

SUMMARY:
The purpose of this study is to determine whether Coronary Computed Tomographic Angiography (CCTA) will increase patient safety by decreasing the rate of missed ACS and adverse events in patients who receive standard care plus CCTA versus standard care alone. Additional goals of the study are to determine whether CCTA can safely reduce the duration of ED visits and the number and duration of hospital admissions.

DETAILED DESCRIPTION:
Justification:

Acute coronary syndrome (ACS) is the clinical manifestation of acute myocardial ischemia induced by coronary artery disease (CAD). Although most patients presenting with chest pain to the Emergency Department (ED) can be stratified into "high risk" or "low risk" chest pain algorithms, patients at "intermediate risk" are more difficult to manage. This translates into lengthy waits in the ED and repetitive investigations while 5.3% of cases of ACS are still missed and too many patients are admitted to the CCU (false positive rate of 14%). CCTA is a novel, non-invasive method for evaluating coronary artery stenosis and occlusion.

The ability to accurately diagnose or exclude ACS in patients in a rapid, non-invasive fashion has been previously lacking. If CCTA is shown to be clinically useful in risk stratification of this patient population, there is great potential for increasing patient safety, reducing ED admission times and decreasing the number and duration of CCU admission.

Objectives:

ED admission and discharge times, CCU consult and decision times and duration of CCU admission, cardiac risk factors, vital signs, laboratory results, ED disposition plan, CCTA results, coronary calcium score, index hospitalization diagnosis, investigations, revascularization rates as well as 30-day diagnosis, death, adverse event rate and subsequent investigations.

Research Method:

The study population will consist of ED chest pain patients at intermediate risk of ACS. Informed consent will be obtained for both CCTA and the 30-day follow up. Patients will be randomized into one of two diagnostic arms: standard care plus CCTA versus standard care alone. If the patient receives CCTA, the test will be interpreted by a blinded radiologist and the results provided to the ED physician and entered into the patient chart. A research nurse will collect workflow and clinical data for all enrolled patients.

Two reviewers, an ED physician and a cardiologist, blinded to the CCTA results, will independently review the index and 30 day clinical data. One of the following will be assigned: acute myocardial infarction, definite unstable angina, possible unstable angina, or no acute coronary syndrome. Alternate non-ACS diagnoses will be ascertained when applicable.

Statistical Analysis This proposal represents a pilot study to demonstrate the feasibility of identifying and recruiting patients to the trial, demonstrate the feasibility of collecting follow-up data, and provide preliminary estimates of outcome measures to help determine the sample size required for a definitive study. All analyses will be descriptive. Recruitment, crossover, follow-up, and completion rates will be determined. Estimates of diagnostic accuracy and length of stay in the ED will be determined and will be used to inform the design of the definitive study.

ELIGIBILITY:
Inclusion criteria (all of the following):

* Anterior or lateral chest pain
* 19 years of age or older
* Fixed address in British Columbia
* Available for telephone follow-up

Exclusion criteria (any of the following).

* Low Risk for ACS (all of the following):
* Age < 40 years with normal ECG (T wave flattening is the only acceptable abnormality)
* No prior history of ischemic chest pain (defined as a past diagnosis of MI or angina, previously prescribed nitroglycerine or a clear history of effort related angina)
* High Risk for ACS (any of the following):
* Diagnosis consistent with ST elevation myocardial infarction
* New ST depression ≥ 0.05 mV
* Troponin > 0.1
* Patients with Killip class III or IV heart failure.
* Hemodynamic instability
* Previous enrolment in this study.
* Presence of terminal noncardiac illness.
* History of angioplasty with stenting and/or grafts.
* Presence of atrial fibrillation.
* Contraindication to administration of iodinated contrast agent.
* Contraindication to beta-blocker administration (eg, asthmatics) AND calcium channel blocker administration.
* Glomerular filtration rate less than 60 mL/min.
* Previous ECG-gated CT with calcium score >1000 Agatston Units.
* Pregnancy.
* Patients with communication difficulties.
* Patients who have a clear alternative diagnosis other than ischemic chest pain (e.g. traumatic chest pain or pneumonia).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2007-11; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
Emergency Department Admission Time | During initial presentation to hospital

SECONDARY OUTCOMES:
CCU consult time | During initial presentation to hospital
CCU decision time | During initial presentation to hospital
Duration of CCU admission | During initial presentation to hospital
Adverse event rate | 30 days post ED visit
All-cause mortality | 30 days post-ED visit

CONTACTS AND LOCATIONS:
Overall Officials: William F Dick, MD, Principal Investigator — Vancouver General Hospital; John Mayo, MD, Study Director — Vancouver General Hospital
Locations (1):
- VGH, Vancouver, British Columbia, Canada